CLINICAL TRIAL: NCT04899336
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Phase 3 Study to Assess the Efficacy, Safety And Immunogenicity of Vaccination With ExPEC9V in the Prevention of Invasive Extraintestinal Pathogenic Escherichia Coli Disease in Adults Aged 60 Years And Older With a History of Urinary Tract Infection in the Past 2 Years
Brief Title: A Study of Vaccination With 9-valent Extraintestinal Pathogenic Escherichia Coli Vaccine (ExPEC9V) in the Prevention of Invasive Extraintestinal Pathogenic Escherichia Coli Disease in Adults Aged 60 Years And Older With a History of Urinary Tract Infection in the Past 2 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109000; VAC52416BAC3001 (Other: Janssen Research & Development, LLC); 2020-005273-27 (EudraCT Number); 2023-506589-30-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Invasive Extraintestinal Pathogenic Escherichia Coli Disease (IED) Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ExPEC9V (Experimental): Participants will receive a single intramuscular (IM) injection of 9-valent extraintestinal pathogenic Escherichia coli vaccine (ExPEC9V) on Day 1.
  Interventions: Biological: ExPEC9V
- Placebo (Placebo Comparator): Participants will receive a single IM injection of matching placebo on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ExPEC9V — ExPEC9V will be administered as an IM injection.
  Other Names: VAC52416,; JNJ-78901563
  Arms: ExPEC9V
Other: Placebo — Matching placebo will be administered as an IM injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of 9-valent extraintestinal pathogenic Escherichia coli vaccine (ExPEC9V) compared to placebo in the prevention of the first invasive extraintestinal pathogenic Escherichia coli disease (IED) event caused by ExPEC9V O-serotypes.

DETAILED DESCRIPTION:
Invasive extraintestinal pathogenic Escherichia coli disease (IED) is defined as an acute illness consistent with systemic bacterial infection, which is microbiologically confirmed either by the isolation and identification of Escherichia coli (E. coli) from blood or any other sterile body sites, or by the isolation and identification of E. coli from urine in a participant with urosepsis and no other identifiable source of infection. ExPEC9V (JNJ-78901563, primary compound number: VAC52416) is a 9-valent vaccine candidate in development for active immunization for the prevention of IED in adults 60 years of age and older. Although IED affects all ages, adults aged greater than or equal to (>=) 60 years have an increased risk of developing IED, including bacteremia and sepsis, which can be community-acquired, hospital-acquired or healthcare associated. As the mechanism of action of conjugate vaccines in the prevention of invasive disease is not expected to be affected by antibiotic resistance mechanisms, that is, resistance mechanisms are not linked to O-polysaccharide structures, the sponsor has no reason to expect a difference in outcome of efficacy between antimicrobial-resistant and susceptible O-serotypes. This study incorporates an inferentially seamless group-sequential design. This study consists of a Screening Phase (selected screening procedures may be performed up to 8 days prior to vaccination on Day 1), Randomization, Vaccination Phase (Day 1) and Follow-up Phase (up to 4 years post-vaccination). The total study duration is approximately up to 6 years 9 months. Key safety assessments include serious adverse events (SAEs), solicited and unsolicited adverse events (AEs), physical examination, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing to share relevant medical information pertaining to medical history and to share medical records relevant to the medical events identified as suspected cases of invasive extraintestinal pathogenic Escherichia coli disease (IED), urinary tract infections (UTI), or acute bacterial prostatitis (ABP) occurring during the study observation period
* Participant must have a history of UTI in the past 2 years for which evidence of diagnosis was verified by the investigator. In case of a recent history of UTI or ABP, the condition must have resolved greater than (>)14 days prior to randomization
* Before randomization, participants who were born female must be either postmenopausal or permanently sterile, and not intending to conceive by any methods
* Participant must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has end-stage renal disease for which dialysis is required
* Participant has a contraindication to intramuscular (IM) injections and blood draws example, due to bleeding disorders or a history of difficult blood draws
* Participant has a history of acute polyneuropathy (for example, Guillain-Barre syndrome) or chronic inflammatory demyelinating polyneuropathy
* Participant has received any Escherichia coli (E. coli) or extraintestinal pathogenic Escherichia coli (ExPEC) vaccine

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17935 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with First Invasive Extraintestinal Pathogenic E.coli Disease (IED) Event with Microbiological Confirmation in Blood or Other Sterile Sites Caused by 9-valent Extraintestinal Pathogenic E. coli Vaccine (ExPEC9V) O-serotypes | Up to 4 years
  Number of participants with first IED event with microbiological confirmation in blood or other sterile sites, excluding IED cases with microbiological confirmation from urine only, caused by ExPEC9V O-serotypes will be reported.

SECONDARY OUTCOMES:
Number of Participants with First IED Event with Microbiological Confirmation in Blood, Other Sterile Sites, or Urine, Caused by ExPEC9V O-serotypes | Up to 4 years
  Number of participants with first IED event, with microbiological confirmation in blood, other sterile sites, or urine, caused by ExPEC9V O-serotypes will be reported.
Number of All IEDs (Including Multiple IEDs per Participant) Caused by ExPEC9V O-serotypes | Up to 4 years
  Number of all IEDs (including multiple IEDs per participant) caused by ExPEC9V O-serotypes will be reported.
Number of Participants with First Hospitalized IED Event Caused by ExPEC9V O-serotypes | Up to 4 years
  Number of participants with first hospitalized IED event caused by ExPEC9V O-serotypes will be reported.
Number of Participants with First IED Event Meeting Criteria for Sepsis Caused by ExPEC9V O-serotypes | Up to 4 years
  Number of participants with first IED event meeting criteria for sepsis caused by ExPEC9V O-serotypes will be reported.
Number of Participants with First Bacteremic IED Event Caused by ExPEC9V O-serotypes | Up to 4 years
  Number of participants with first bacteremic IED event caused by ExPEC9V O-serotypes will be reported.
Number of Participants with First Pyelonephritis Event Caused by ExPEC9V O-serotypes | Up to 4 years
  Number of participants with first pyelonephritis event caused by ExPEC9V O-serotypes will be reported.
Number of Participants with First Urinary Tract Infection (UTI) Event Caused by ExPEC9V O-serotypes | Up to 3 years
  Number of participants with first UTI event caused by ExPEC9V O-serotypes will be reported.
Number of All UTIs (Including Multiple UTIs per Participant) Caused by ExPEC9V O-serotypes | Up to 3 years
  Number of all UTIs (including multiple UTIs per participant) caused by ExPEC9V O-serotypes will be reported.
Number of Participants with First IED Event Caused by Escherichia coli (E.coli) | Up to 4 years
  Number of participants with first IED event caused by E.coli will be reported.
Number of Participants with First Pyelonephritis Event caused By E.coli | Up to 4 years
  Number of participants with first pyelonephritis event caused by E.coli will be reported.
Number of Participants with First UTI Event caused by E.coli | Up to 3 years
  Number of participants with first UTI event caused by E.coli will be reported.
Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex Electrochemiluminescent (ECL)-based Immunoassay | Up to 4 years
  Antibody titers to vaccine O-serotype antigens as determined by multiplex ECL-based immunoassay will be reported.
Antibody Titers to Genetically Detoxified Form of Exotoxin A Derived from Pseudomonas Aeruginosa (EPA) as Determined by Multiplex ECL-based Immunoassay | Up to 4 years
  Antibody titers to EPA as determined by multiplex ECL-based immunoassay will be reported.
Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex Opsonophagocytic Assay (MOPA) | Up to 4 years
  Antibody titers to vaccine O-serotype antigens as determined by MOPA will be reported.
Number of Participants with Solicited Local Adverse Events (AEs) | Up to Day 15 (until 14 days post-vaccination)
  Number of participants with solicited local AEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs are pre-defined local (at the injection site) AEs. Participants will be asked to note in the diary occurrences of injection site pain/tenderness, erythema and swelling at the study vaccine injection site daily for 14 days post-vaccination (day of vaccination and the subsequent 14 days).
Number of Participants with Solicited Systemic AEs | Up to Day 15 (until 14 days post-vaccination)
  Number of participants with solicited systemic AEs will be reported. Participants will be instructed on how to record daily temperature using a thermometer and also instructed to note signs and symptoms in the diary on a daily basis for 14 days post-vaccination (day of vaccination and the subsequent 14 days). Solicited systemic AEs are fatigue, headache, nausea, and myalgia.
Number of Participants with Unsolicited AEs | Up to Day 30 (until 29 days post-vaccination)
  Number of participants with unsolicited AEs will be reported. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Number of Participants with Serious Adverse Events (SAEs) | Up to 181 days
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with SAEs Related to Study Vaccine or Study Procedures | Up to 4 years
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important. Participants with SAEs related to study procedures or vaccines will be reported in this outcome measure.
Short Form-36 (SF-36) Total Scores | Up to 4 years
  The SF-36 is a 36-item questionnaire with a recall period for all items of 1 week. The SF 36 version 2 includes 8 domains that measure physical functioning, role limitations due to physical health problems, bodily pain, general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE) and mental health (MH). The 8 domains can be aggregated into 2 summary scales that reflect physical and mental health: a physical component summary (PCS) and a mental component summary (MCS). Responses to all items are rated on a 3-, 5- or 6-point Likert scale. The scores range from 0 (lowest or worst possible level of functioning) to 100 (highest or best possible level of functioning).
European Quality of Life (EuroQol) 5-Dimension 5-Level Questionnaire (EQ-5D-5L) Scores | Up to 4 years
  The EQ-5D-5L is a standardized measure of health status. It is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in Frailty Index | Baseline to 4 years
  Frailty will be assessed at baseline based on Short Physical Performance Battery (SPPB) score and will be calculated using participants self-reported information regarding health status (components of SF-36 and EQ-5D), and baseline health conditions collected through medical conditions of interest. The specific medical conditions of interest used for the calculation of the frailty index score will include: diabetes mellitus, history of myocardial infarction, congestive heart failure, hypertension, history of cerebrovascular disease (sequelae of stroke), chronic obstructive pulmonary disease (COPD), cancer, osteoarthritis or rheumatoid arthritis, gastric or duodenal ulcer, long term disability or handicap, hearing problems, migraine, cataract, and glaucoma. Total Frailty Index, ranging from 0 (not frail or best possible score) to 43 (frail or worst possible score), will be calculated as accumulation of individual's deficits.
Medical Resource Utilization (MRU) for IED Events Caused by ExPEC9V O-Serotype | Up to Day 366 Post-IED
  MRU for IED events caused by ExPEC9V O-serotype will be reported.
MRU for UTI Events Caused by ExPEC9V O-Serotype | Up to Day 29 Post-UTI
  MRU for UTI events caused by ExPEC9V O-serotype (for immunogenicity subset only that is for participants from selected study sites who have given informed consent prior to randomization for additional immunogenicity assessments) will be reported.
MRU for Acute Bacterial Prostatitis (ABP) Events Caused by ExPEC9V O-Serotype | Up to Day 29 Post-ABP
  Medical resource utilization for ABP events caused by ExPEC9V O-serotype (for immunogenicity subset only that is for participants from selected study sites who have given informed consent prior to randomization for additional immunogenicity assessments) will be reported.
Number of Participants with the Hospitalization for IED or, UTI, or ABP Events Caused by ExPEC9V O-Serotype | Up to 4 years
  Number of participants with hospitalization for IED or, UTI, or ABP events caused by ExPEC9V O-serotype will be reported.
Length of Stay in Hospital for IED, UTI, or ABP Events Caused by ExPEC9V O-Serotype | Up to 4 years
  Length of stay in hospital for IED, UTI, or ABP events caused by ExPEC9V O-serotype will be reported.
Number of Participants with the Intensive Care Unit (ICU) Hospitalization for IED or UTI or ABP Events Caused by ExPEC9V O-Serotype | Up to 3 months post clinical event
  Number of participants with ICU hospitalization for IED or UTI or ABP events caused by ExPEC9V O-serotype will be reported.
Length of ICU Stay in Hospital for IED, UTI, or ABP Events Caused by ExPEC9V O-Serotype | Up to 3 months post clinical event
  Length of ICU stay in hospital for IED, UTI, or ABP events caused by ExPEC9V O-serotype will be reported.
Number of Participants with IED-related and All-cause Mortality | Up to 4 years
  Number of participants with IED-related and all-cause mortality will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (372):
- United States (141):
  - Lakeview Clinical Research, Guntersville, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - Interspond-Clinical Research Institute of AZ, Sun City West, Arizona
  - Baptist Health Center For Clinical Research, Little Rock, Arkansas
  - Sun Urology - Buena Park Office, Buena Park, California
  - Hope clinical Research LLC, Canoga Park, California
  - Velocity Clinical Research, Inc., Chula Vista, California
  - Marvel Clinical Research, Huntington Beach, California
  - California Adult Circumcision - Alvarado La Mesa Urology Center, La Mesa, California
  - Om Research LLC, Lancaster, California
  - Atlantic Urology Medical Group, Long Beach, California
  - Long Beach Clinical Trials, LLC, Long Beach, California
  - American Institute of Research, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Comprehensive Urology, Los Angeles, California
  - Veterans Affairs Greater Los Angeles HCS, Los Angeles, California
  - VA Sacramento Medical Center, Mather, California
  - Hoag Medical Group, Newport Beach, California
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - Empire Clinical Research, LLC, Pomona, California
  - Inland Urology Medical Group, Pomona, California
  - UC Davis Health System, Sacramento, California
  - Northern California Research, Sacramento, California
  - San Diego Sports Medicine & Family Health Center, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - California Kidney Specialists, San Dimas, California
  - Prestige Medical Group, Santa Ana, California
  - Millennium Clinical Trials LLC, Simi Valley, California
  - San Antonio Regional Hospital, Upland, California
  - Yale University, New Haven, Connecticut
  - Ideal Clinical Research, Adventura, Florida
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Clinical Research of Brandon, Brandon, Florida
  - Moore Clinical Reseach - Brandon Clinic, Brandon, Florida
  - Florida Medical Center of Clearwater, Clearwater, Florida
  - Innovative Research of West Florida, Incorporated, Clearwater, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Prestige Clinical Research Center, Inc., Coral Gables, Florida
  - Accel Research Sites, DeLand, Florida
  - Doral Medical Research, Doral, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - Indago Research & Health Center Inc, Hialeah, Florida
  - Prestige Clinical Research, Homestead, Florida
  - Multi Specialty Research Associates Inc, Lake City, Florida
  - ClinCloud Clinical Research, Maitland, Florida
  - Nova Clinical Research Center, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Royal Care Medical Research Corporation, Miami, Florida
  - Retreat Medical Research LLC, Miami, Florida
  - Suncoast Research Group, Miami, Florida
  - Continental Research, Miami, Florida
  - Dynamic Medical Research, LLC, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - Health- Life Research Inst, Miami, Florida
  - Office of Dr. Marisela Gonzalez, Miami, Florida
  - Felicidad Medical Research, Miami, Florida
  - A and R Research Group, Miami, Florida
  - Alpha Science Research, Miami, Florida
  - Clinical NeuroScience Solutions Inc, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - Pines Care Research Center Inc, Pembroke Pines, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Care Access Research, Spring Hill, Florida
  - Tampa General Hospital, Tampa, Florida
  - Theia Clincial Research, LLC, Tampa, Florida
  - Precision Research Institute, Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Care Access Research, Tampa, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Northwestern Medicine - Northwestern Memorial Hospital Galter Pavilion, Chicago, Illinois
  - Jesse Brown VAMC Department of Surgery, Chicago, Illinois
  - University Of Illinois, Chicago, Illinois
  - Medisphere Medical Research Center, Llc, Evansville, Indiana
  - Asha Clinical Research-Munster Llc, Hammond, Indiana
  - Mishawaka Osteopathic Clinic/MOC Research, Mishawaka, Indiana
  - Cypress Medical Research Center, Wichita, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - KAMP Medical Research, Inc, Natchitoches, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Kaiser Permanente, Rockville, Maryland
  - Floating Hospital For Children at Tufts Medical Center, Boston, Massachusetts
  - West Roxbury Veterans Affairs Medical Center, West Roxbury, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - MediSync Clinical Research, Petal, Mississippi
  - Meridian Clinical Research, LLC, Grand Island, Nebraska
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Hope Research Institute, Las Vegas, Nevada
  - Sierra Clinical Research, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - I.D. Care, Inc., Hillsborough, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Meridian Clinical Research, LLC, Binghamton, New York
  - Meridian Clinical Research, LLC, Endwell, New York
  - Manhattan Medical Research, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Durham VAMC, Durham, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - ECU Health Vidant Medical Center, Greenville, North Carolina
  - Plains Clinical Research, Fargo, North Dakota
  - Kroger Health, Centerville, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - Kroger Health, Englewood, Ohio
  - The Little Clinic, Englewood, Ohio
  - Comprehensive Internal Medicine, Wooster, Ohio
  - Tekton Research Inc., Yukon, Oklahoma
  - Kaiser Permanente, Portland, Oregon
  - Capital Area Research, Camp Hill, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Hugh D. Durrence, MD, PC, Charleston, South Carolina
  - Waterway Familiy Medicine, Little River, South Carolina
  - Novel Research LLC, Bellaire, Texas
  - Global Medical Research - Dallas, Dallas, Texas
  - Medical City Dallas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Digestive Health Associates, Houston, Texas
  - EPIC Clinical Research, Lewisville, Texas
  - SMS Clinical Research LLC, Mesquite, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Audie L Murphy Memorial Va Ho, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Lone Peak Family Medicine, Draper, Utah
  - Clinical Alliance for Research and Education, Annandale, Virginia
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Infectious Disease Associates of Central Virginia, Lynchburg, Virginia
  - IACT - Suffolk Multispecialty Research, Suffolk, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Multicare Institute For Research & Innovation - Rockwood Clinic - Cheney, Cheney, Washington
  - Exemplar Research, Inc, Morgantown, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Australia (14):
  - Saint Andrew's War Memorial Hospital, Brisbane
  - GP Surgery - Campbelltown, Campbelltown
  - Barwon Health - University Hospital Geelong, Geelong
  - CMAX Clinical Research, Melbourne
  - John Hunter Hospital, New Lambton
  - Fiona Stanley Hospital, Palmyra DC
  - McIntyre Medical Center, Para Hills West
  - North West Medical Center, Salisbury
  - Mater Medical Centre South Brisbane, South Brisbane
  - Bene Aged Care - Italian Village, St Agnes
  - Westmead Hospital, Sydney
  - AusTrials Pty Ltd, Taringa
  - AusTrials Pty Ltd, Tarragindi
  - Adelaide Medical Solutions, Woodville
- Canada (9):
  - CARe Clinical Ltd, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - CARe Clinical Ltd, Red Deer, Alberta
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - Health Sciences North, Greater Sudbury, Ontario
  - Dawson Road Family Health Team, Guelph, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - Alpha Recherche Clinique, Québec, Quebec
- China (13):
  - West China School of Medicine/West China Hospital, Sichuan University, Chengdu
  - Funan Center for Disease Control and Prevention, Fuyang
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - 1st Affiliated Hospital of Zhejiang University Medical College, Hangzhou
  - Anhui Provincial Center for Disease Control and Prevention, Hefei
  - Huoqiu County Center For Disease Control and Prevention, Liuan
  - Jiangsu Provincial Center for Disease Control and Prevention, Nanjing
  - Nanjing Medical University, Nanjing
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Suzhou Municipal Hospital, Suzhou
  - Taizhou Peoples Hospital, Taizhou
  - Yixing People's Hospital, Wuxi
- Colombia (11):
  - Clinica de la Costa, Barranquilla
  - IPS Centro Cientifico Asisitencial Jose Luis Accini S.A.S., Barranquilla
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED, Casanare
  - Fundacion Cardiovascular de Colombia, Floridablanca
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED, Girardot
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED, Helechos
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
  - CAIMED Acacias, Meta
  - Fundacion Centro de Investigaciones Clinicas IPS Cardiomet, Pereira
  - Corporación Clínica Universidad Cooperativa De Colombia Clínica Ucc, Villavicencio
- Czechia (13):
  - Uromeda, Brno
  - Ordinace Hradebni s.r.o., České Budějovice
  - Aesculap Ambulance sro - Zdravotni Stredisko Centrum Zdravi, Dolní Břežany
  - Centrum Ockovani a Cestovi Mediciny, Hradec Králové
  - Res Medica, Nový Knín
  - PreventaMed, s.r.o., Olomouc
  - GYNURO s.r.o, Ostrava-Proskovice
  - Ambulance name: Gynekologická ordinace MUDr, Pilsen
  - MUDr. Mita Rosenberg, Pilsen
  - Gona s.R.o- Orfinace Harov, Prague
  - Zdravi-fit, s.r.o., Protivín
  - Nemocnice Slany, Slaný
  - Progerint s.r.o., Vysoké Mýto
- Denmark (6):
  - Aalborg Universitetshospital Nord, Hellerup
  - Gentofte Hospital, Herlev
  - Nordsjaellands Hospital - Hillerod, Hilleroed
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense M
  - Sjællands University hospital, Roskilde
- France (7):
  - Centre Hospitalier Annecy Genevois, Annecy
  - CHU Dijon Bourgogne - Hopital Francois Mitterrand, Dijon
  - CHU de Limoges, Limousis
  - Hopital de La Croix Rousse, Lyon
  - CHU Nimes Hopital Caremeau, Nîmes
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
- Germany (8):
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitatsklinikum Jena, Jena
  - Familienmedizinisches Zentrum Radowsky, Leipzig
  - SIBAmed GmbH & Co. KG, Leipzig
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Red-Institut für medizinische Forschung und Fortbildung, Oldenburg in Holstein
  - Praxis Dr. Weimer, Reinfeld
  - Universitaetsmedizin Rostock, Rostock
- India (10):
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre (MRC), Belagavi
  - S. R. Kalla Memorial General Hospital, Jaipur
  - Nil Ratan Sircar Medical College and Hospital, Kolkata
  - Regency health super specialty hospital, Lucknow
  - Asian Institute Of Medical Science, Mumbai
  - Jagadguru Sri Shivarathreeshwara Academy of Higher Education and Research, Mysuru
  - Indraprastha Apollo Hospital, New Delhi
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Nirmal Hospital Pvt. Ltd., Surat
  - BAPS Pramukhswami Hospital, Surat
- Israel (5):
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - ASL2 Lanciano - Vasto - Chieti - Ospedale 'SS Annunziata' di Chieti, Chieti
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera Sant Andrea, Rome
- Japan (32):
  - Akashi Medical Center, Akashi Shi
  - Fukuoka Shinmizumaki Hospital, Fukuoka
  - Fukuoka Wajiro Hospital, Fukuoka
  - Hakodate Goryoukaku Hospital, Hakodate
  - Matsunami General Hospital, Hashima-gun
  - Teine Keijinkai Hospital, Hokkaido
  - Aso Co.,Ltd Iizuka Hospital, Iizuka
  - Inoue Hospital, Itoshima
  - Kano Hospital, Kasuya-gun
  - Kanto Rosai Hospital, Kawasaki
  - Shinkomonji hospital, Kitakyushu
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu
  - JRC Nagasaki Genbaku Hospital, Nagasaki
  - Kyoujinkai Clinic Komatsu, Neyagawa
  - Omuta City Hospital, Omuta-Shi
  - Kyobashi Sugimoto Clinic, Osaka
  - Japan Community Health Care Organization Osaka Hospital, Osaka
  - Abe Diabetes Clinic, Ōita
  - Almeida Memorial Hospital, Ōita
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - National Hospital Organization Shikoku Cancer Center, Sanuki
  - Teine Maeda Urology Clinic, Sapporo
  - Teine Urological Clinic, Sapporo
  - Nanbu Tokushukai Hospital, Shimajiri-Gun
  - Shimonoseki City Hospital, Shimonoseki-shi
  - Tokyo Shinagawa Hospital, Shinagawa City
  - Suita Tokushukai Hospital, Suita-Shi
  - Japanese Red Cross Society Suwa Hospital, Suwa-Shi
  - Japan Community Health care Organization Kyushu Hospital, Yahatanishi-ku
  - Shimonoseki City Hospital, Yamaguchi
  - Yokohama Rosai Hospital, Yokohama
  - National Hospital Organization Yokohama Medical Center, Yokohama
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - Ziekenhuis, Uden
  - The Julius Center - Utrecht Science Park - Stratenum, Utrecht
- New Zealand (20):
  - Southern Clinical Trials Totara Clinical Research, Auckland
  - Southern Clinical Trials Ltd, Auckland
  - Optimal Clinical Trials, Auckland
  - Tauranga Urology Research Limited, Bay of Plenty
  - Canterbury Urology Research Trust, Christchurch
  - Southern Clinical Trials Ltd, Christchurch Central
  - P3 Research Ltd, Dunedin
  - Lakeland Clinical Trials, Hamilton
  - P3 Research Ltd, Hastings
  - P3 Research - Lower Hutt, Lower Hutt
  - Southern Clinical Trials Ltd, Nelson
  - P3 Research Ltd, Palmerston North
  - Culloden Research Ltd, Papamoa
  - Middlemore Clinical Trials, Papatoetoe
  - Optimal Clinical Trials, Rosedale
  - Lakeland Clinical Trials, Rotorua
  - P3 Research Ltd, Tauranga
  - Lakeland Clinical Trials, Upper Hutt
  - P3 Research Limited Kapiti, Wellington
  - Capatial & Coast District Health Board, Wellington
- South Korea (15):
  - Dong-A University Hospital, Busan
  - Hallym University Chuncehon Medical Center, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Chunnam National University Hospital, Gwangju
  - Korea University Ansan Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Hallym University Sacred Heart Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic university of Korea, St. Vincent's Hospital, Suwon
  - WonJu Severance Christian Hospital, Wŏnju
- Spain (19):
  - Hosp. Gral. Univ. Dr. Balmis, Alicante
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. de Bellvitge, Barcelona
  - Hosp. Del Mar, Barcelona
  - Consorci D'Atenció Primària de Salut Barcelona Esquerra, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - CAP Dr. Vicenç Papaceit ABS LA ROCA, La Roca del Vallès
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hospital Sanitas La Moraleja, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp. Quirónsalud Málaga, Málaga
  - Complexo Hosp. Univ. de Ourense, Ourense
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Virgen Macarena, Seville
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (8):
  - Helsingborgs lasarett, Helsingborg
  - BTH Research & Development Clinic, Karlskrona
  - CTC Ebbepark, Linkoaping
  - Skanes universitetssjukhus, Malmo
  - CTC GoCo, Mölndal
  - Universitetssjukhuset Orebro, Örebro
  - ClinSmart Sweden AB, Solna
  - ClinSmart Sweden AB, Uppsala
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Thailand (5):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Thai Red Cross Aids Research Centre, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Tropical Medicine Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
- United Kingdom (27):
  - Aberdeen Royal Infirmary, Aberdeen
  - Atherstone Surgery, Atherstone
  - Banbury Cross Health Center, Banbury
  - FutureMeds Bridle Clinic, Birkenhead
  - FutureMeds-Soho UK, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - North Bristol NHS Trust, Bristol
  - University Hospitals Bristol NHS Trust, Bristol
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Eynsham Medical Centre, Eynsham
  - The Garth Surgery, Guisborough
  - University Hospitals Of Leicester Nhs Trust, Leicester
  - King's College Hospital NHS Foundation Trust, London
  - Manchester Royal Infirmary, Manchester
  - The NIHR Manchester Clinical Research Facility, Manchester
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Plymouth University Hospitals Trust, Plymouth
  - Ashgrove Surgery, Pontypridd
  - The Adam Practice, Poole
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Midlands Partnership NHS Foundation Trust, Stafford
  - North Tees Furturemeds, Stockton-on-Tees
  - Mid Yorkshire Hospital NHS Trust- Pinderfields Hospital, Wakefield
  - Church Street Practice, Wantage
  - Windrush Medical Practice, Witney

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Doua J, Ekkelenkamp M, Verheij T, Go O, Ruhmel S, Leathers K, Spiessens B, van Rooij S, Fowler VG Jr, Geurtsen J, Dolor R, Sarnecki M, Chatterjee R, Poolman J, Bonten M; on behalf COMBACTE-NET consortium/EXPECT study group. Feasibility of tracking invasive Escherichia coli disease among older adults in a community setting: A prospective observational study. Eur J Clin Microbiol Infect Dis. 2024 Mar;43(3):541-550. doi: 10.1007/s10096-023-04738-y. Epub 2024 Jan 18. PMID 38236365